CLINICAL TRIAL: NCT04859205
Title: The SUPPORT-Pro Online Platform: Helping Healthcare Professionals to Increase Their Confidence Levels in Treating Individuals Living With T1D
Brief Title: The SUPPORT-Pro Online Platform for Healthcare Professionals Treating Individuals Living With T1D
Acronym: SUPPORT-Pro
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Institut de Recherches Cliniques de Montreal (Other)
Responsible Party: Principal Investigator, Anne-Sophie Brazeau, Associate Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-1107
Record Dates: First submitted 2021-04-12; First posted 2021-04-26 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Educational Activities
Keywords: Type 1 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Methods

STUDY DESIGN:
Intervention Model Description: This study is a non-randomized pre-post trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention (Experimental): All participants partaking the SUPPORT-Pro study will receive the full intervention for 3 months which implies: (1) Full access to the platform (2) a newsletter sent by email every 2 weeks to inform them on the new blogs posted on the platform.
  During the following 9 months, participants will still have access to the platform, but no newsletter will be sent (sustainability phase).
  Interventions: Behavioral: Intervention

INTERVENTIONS:
Behavioral: Intervention — Participants will have access to the SUPPORT-Pro self-guided online training platform addressing many aspects of type 1 diabetes care. The SUPPORT-Pro content was developped by a team of health professionals specialized in type 1 diabetes as well as patient partners. It's content is regularly updated, evidence-based and divided into 6 categories (medication, blood glucose monitoring, diet, physical activity, hypo and hyperglycemia, health and other particularities). In each category, users can pick between 3 levels (beginner, intermediate and advanced) according to their level of confidence and knowledge.
  Participants will be asked to fill out questionnaires at baseline, 3-month, and 12-month of the intervention which include the following: Eligibility assessment, identification, background, confidence, platform satisfaction.

SUMMARY:
Health care professionals (HCPs) help an support patients living with type 1 diabetes (PWT1D) who need to achieve optimal blood glucose control in order to prevent short and long term complications of T1D. However, studies show that not all HCPs are aware of T1D management as most of them only see PWT1D occasionally. This makes it difficult for HCPs to remain aware of the particularities of the condition and stay up-to-date on rapidly evolving technologies and therapies available. Moreover, low confidence levels and the inaccessibility to continuing medical education on the specificities of new therapies and technologies might increase the failure of HCPs to propose the optimal treatment plan to their PWT1D.

The SUPPORT online platform, that was first developed for PWT1D, was adjusted to suit the needs of HCPs (SUPPORT-Pro). The regularly updated bilingual (English and French) peer-reviewed content of SUPPORT, which covers the various elements that an individual with T1D needs to know to manage the disease and aims at making a better use of technologies and new therapies, is the first in its kind and is highly relevant for HCPs.

The main objective of this study is to determine if the SUPPORT-Pro online training platform can increase HCPs' (dietitians, nurses, pharmacists, medical doctors) confidence level in treating individuals with T1D. This study is a non-randomized pre-post trial. We hypothesize that the training provided through the SUPPORT-Pro online platform will significantly increase HCPs' confidence level in treating individuals with T1D after 3 months when compared to their confidence level before the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Certified Health Care Professional (nurse, physician (including resident in medicine), dietitian, pharmacist) who is member of a regulatory body in Canada
2. Self-reported working with at least 1 patient with type 1 diabetes in the last six months
3. Has access to the Internet
4. Use of an active email address
5. Comprehension of English or French

Exclusion Criteria:

1. Certified diabetes educators
2. Working in a T1D specialized clinic
3. Living with T1D
4. Currently living with someone with T1D (e.g. kid, partner, etc.)
5. Working in the pharmaceutical industry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
To compare the level of confidence in treating individuals with type 1 diabetes measured at 3 months to the level of confidence measured at baseline. | 3 months
  Levels of confidence will be measured using a questionnaire inspired from the Maternal Self-Efficacy for Diabetes Management Scale (MSED). For this study, MSED was modified to better assess the self-confidence of health care professionals. We have converted the 17-item questionnaire to a 19-item questionnaire (removing questions specific to familial support and adding questions on new therapies and technologies) and edited the wording of the questions. Every item is rated on a scale from 1 to 5. The satisfaction score will be the sum of all items, on a maximum of 95.
  Confidence levels at 3 months and at baseline will be compared using paired t-test with a 95% confidence interval, if normality assumption of the paired difference holds. Otherwise, the non-parametric counterpart, Wilcoxon signed-rank test, will be used and a 95% non-parametric confidence interval will be provided.

SECONDARY OUTCOMES:
To compare, in each specific group of HCPs (nurses, dietitians, doctors and pharmacists), the confidence levels in treating their patients with T1D after 3 months of access to the SUPPORT-Pro platform with confidence at baseline. | 3 months
  Levels of confidence will be measured using a questionnaire inspired from the Maternal Self-Efficacy for Diabetes Management Scale (MSED). For this study, MSED was modified to better assess the self-confidence of health care professionals. We have converted the 17-item questionnaire to a 19-item questionnaire (removing questions specific to familial support and adding questions on new therapies and technologies) and edited the wording of the questions. Every item is rated on a scale from 1 to 5. The satisfaction score will be the sum of all items, on a maximum of 95.
  Confidence levels at 3 months and at baseline will be compared using paired t-test with a 95% confidence interval, if normality assumption of the paired difference holds. Otherwise, the non-parametric counterpart, Wilcoxon signed-rank test, will be used and a 95% non-parametric confidence interval will be provided.
To measure the sustainability of change in all HCPs' confidence in treating patients with T1D at 12 months | 12 months
  Levels of confidence will be measured at baseline, after 3 months and after 12 months using a questionnaire inspired from the Maternal Self-Efficacy for Diabetes Management Scale (MSED). For this study, MSED was modified to better assess the self-confidence of health care professionals. We have converted the 17-item questionnaire to a 19-item questionnaire (removing questions specific to familial support and adding questions on new therapies and technologies) and edited the wording of the questions. Every item is rated on a scale from 1 to 5. The satisfaction score will be the sum of all items, on a maximum of 95.
  Sustainability of change will be assessed by comparing level of confidence at the 3 time points using a one-way repeated measures ANCOVA, with change from baseline as the outcome, and baseline level of confidence adjusted for in the model.
Time spent on the platform | 3 months
  Using back-end data collected from Google Analytics, the total time (in minutes) spent on the platform during 3 months will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on its normality.
Number of posts of the discussion forum | 3 months
  Using back-end data collected from Google Analytics, the number of posts on the discussion forum forum will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on its normality.
Number of completed courses | 3 months
  Using back-end data collected from Google Analytics, the number of completed courses will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on its normality.
Number of completed categories | 3 months
  Using back-end data collected from Google Analytics, the number completed category (maximum of 6) will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on its normality.
Number of viewed videos | 3 months
  Using back-end data collected from Google Analytics, the number of viewed videos will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on its normality.
Satisfaction of the platform. | 3 months
  After using the platform for 3 months, participants will be invited to complete a satisfaction questionnaire which includes open ended questions and a 7-items Likert scale (from 1 to 7, total score on 49).
  Continuous endpoints will be presented using mean and SD (standard errors) or median and interquartile intervals, depending on their normality. Categorical variables will be presented using frequencies and percentages.

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie Brazeau, PhD, Principal Investigator — McGill University
Locations (1):
- Institut de Recherches Cliniques de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No